CLINICAL TRIAL: NCT03392831
Title: Comparative Cost-Effectiveness and Safety of Infusional Therapy With Central Venous Catheters Versus Peripherally Inserted Central Catheters: a Randomized Clinical Trial
Brief Title: PIcc Cost EffectiveneSS and Safety of Infusional Therapy
Acronym: PrInCESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 170529
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Thrombosis; Infection
Keywords: Central Venous Catheters; Vascular Access Devices; Nursing; Cost Effectiveness; PICC
MeSH Terms: conditions — Thrombosis; Infections | interventions — Catheterization, Peripheral; Central Venous Catheters

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Open Blinded End-Point (PROBE) study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripherally inserted central catheter (Experimental): The peripherally inserted central catheter (PICC) with 3 to 6 French calibers, with one, two or three lumens Groshong and PowerPICC models. These calibers are dependent on the amount of lumens, which are used for single or concomitant infusions.
  Interventions: Other: Peripherally inserted central catheter (PICC)
- Central venous catheter (Active Comparator): The central venous catheter (CVC), with a short stay of 3 to 7 French gauges with one or more lumens.
  Interventions: Other: Central venous catheter

INTERVENTIONS:
Other: Peripherally inserted central catheter (PICC) — The peripherally inserted central catheter with different sizes (French scale). Trained vascular access nurses will perform the insertion of the PICC, guided by ultrasound at bedside using the Seldinger technique. A suitable sterile field will be established. In the case of children the procedure may be performed at the Ambulatory Surgical Center
  Arms: Peripherally inserted central catheter
Other: Central venous catheter — The central venous catheter with different sizes (French scale). Trained doctors will perform the insertion of the CVC, guided by ultrasound at bedside using the Seldinger technique. A suitable sterile field will be established.The decision of the caliber depends on the clinical evaluation and need for multiple infusional therapy.
  Arms: Central venous catheter

SUMMARY:
Infusion therapy comprises the parenteral administration of solutions, through peripheral or central vascular access. Some solutions and drugs are highly irritating to the vascular endothelium and therefore cannot be administered in peripheral vessels, because increase the risk of phlebitis and/or tissue necrosis. Thus, the alternative is the central venous catheter (CVC) where the access can be by direct puncture of a central vessel or peripheral vessel puncture with progression of the catheter until central positioning, through a peripherally inserted central catheter (PICC).

We must take into account that indication, insertion, handling and maintenance must be balanced with risks, benefits and costs. The insertion and maintenance of both catheters are not free of complications. Among the most frequent are: Infection, thrombosis, lumen occlusion and accidental early removal of the catheter. This often implies in the need for new vascular access, impacting on morbidity and increased treatment costs.

The PICC has some advantages over CVC, for example: avoids repetitive punctures and consequently decreased handling/pain; a lower risk of infection; avoids the use of venous dissections; reduces the risks of pneumothorax/hemothorax; reduces the risk of infiltration, extravasation, necrosis tissue and chemical phlebitis. Further, the PICC can be used as a long-term catheter with easy handling in extra-hospital condition. All these advantages suggest that this technology offers lower cost to the health system and more benefits for patients. However, PICC is not available for use in infusion therapy in patients of the Brazilian public health system, except for neonates.

The available literature does not address cost-effectiveness studies of this technology in the international scope comparing the PICC versus CVC. And, similarly, we do not have studies conducted in Brazil to incorporate this technology into our public health system, based on its benefits and potential cost reduction.

In order to fill this gap, this study aims to test if the use of PICC in patients with infusional therapy equal or superior to 10 days (Intervention Group), will show a lower incidence in the outcomes (infection, thrombosis or mechanical complications), besides being more cost-effective when compared to the use of CVC of short stay (Control Group).

DETAILED DESCRIPTION:
Patient recruitment: Adult and pediatric patients will be included during hospitalization in the clinical/surgical units at the Hospital de Clínicas de Porto Alegre.

Variables of registry: Clinical data (diagnosis, reason for indication of catheter, site of insertion, vessel size, pharmacological treatment); Socio-demographic (age, sex, education, income); Ultrasonography (vessel evaluation); Radiography (to ensure the correct positioning of the catheter); economic variables (costs of all inputs used).

Data collection: All variables will be recorded in an instrument developed by the authors.

Statistical analysis: Continuous variables will be described using means and standard deviations or median and range in case of asymmetric distribution of data. Categorical variables will be presented using frequency distribution. Analyses will be conducted using chi-square and t tests for independent samples. P values <0.05 will be considered statistically significant. A Statistical Package for Social Sciences v.20.0 will be used. The Cox Regression Analysis and Log-rank test will compare the groups in relation to complication-free survival.

Cost-effectiveness analysis: The cost-effectiveness analysis will be measured by the incremental cost-effectiveness ratio (ICER), showed by the difference in cost between intervention and control group, divided by the difference in their effect. It represents the average incremental cost associated with 1 additional unit of the measure of effect. The cost-effectiveness analysis will be based on the cost estimate for insertion and maintenance of the catheter, including values of the inputs used, medicines, costs with professionals, surgical environment, laboratory and imaging exams.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 5 years old,
* Hospitalized,
* With prescription of infusion therapy for 10 days or more of antibiotics, antineoplastics or other drugs with a pH lower than 5 or higher than 9 and / or osmolarity above 900 mOsm / l, parenteral nutrition or hypertonic solutions.

Exclusion Criteria:

* Insertion of the central catheter in emergency situations.
* Critical patient in the acute or terminal stage;
* Chronic renal disease stage IV or V and indication of hemodialysis;
* Pediatric patients with leukemia until the induction phase;
* Adult patients diagnosed with acute myeloid leukemia;
* Autologous and allogenic marrow transplantation;
* Upper limb with anatomical alteration, presence of arteriovenous fistula, axillary emptying or previous vascular procedure;
* Presence of skin changes in the area of the puncture, such as thrombophlebitis, dermatitis, cellulitis, burn among others;
* Patient using crutches or devices that require exertion or support in the upper limbs.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 624 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
infectious complications | up to 30 days or the end of therapy
  bloodstream infection
thrombotic complications | up to 30 days or the end of therapy
  radiographically-confirmed upper-extremity deep vein thrombosis
mechanical complications | up to 30 days or the end of therapy
  chest X-ray
accidental removal | up to 30 days or need for another catheter
  obstruction or accidental removal

SECONDARY OUTCOMES:
Cost Effectiveness | up to 30 days or the end of therapy
  reduction of the rates composite outcome of complications
  * Catheter occlusion: significant reduction of infusion flow or an impairment of blood back-flow;
  * Catheter damage, malposition and catheter migration.

CONTACTS AND LOCATIONS:
Overall Officials: Carisi A Polanczyk, Study Director — Federal University of Rio Grande do Sul - Faculty of Medicine; Marco A Lumertz Saffi, Study Director — Hospital de Clinicas de Porto Alegre; Jeruza L Neyeloff, Study Director — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: No